CLINICAL TRIAL: NCT00978094
Title: Validation of a Novel Sham Cervical Spinal Manipulation Procedure.
Status: Completed | Type: Observational
Sponsor: Canadian Memorial Chiropractic College (Other)
Responsible Party: Howard Vernon, Canadian Memorial Chiropractic College
Other Study IDs: 072155; 1R21AT004396-01A1 (NIH)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary hypotheses:

Ho1: In chronic neck pain patients, randomly treated with either a "sham" or "real" cervical manipulation procedure, the probability of perceiving a Real Manipulation Procedure is equal to the probability of obtaining a Real Manipulation Procedure, AND, Ho2: Spinal tenderness will remain unchanged following the treatment procedure for both groups.

Secondary (null) hypotheses:

1. Neck pain, cervical ranges of motion and paraspinal EMG responses to pressure pain will remain unchanged in both groups;
2. there will be no differences between groups with respect to 2a) neck joint cavitations and 2b) forces across the cervical spine measured during the manoeuvres.

DETAILED DESCRIPTION:
1. Develop a randomized controlled clinical trial design to optimize the testing of the effects of a sham vs real cervical manipulation.
2. Use novel modifications of both a sham a real manipulation to create "procedures" designed to optimize group equivalence in the RCT design. Then, evaluate the accuracy of 'patient post-treatment perception of treatment type' versus actual administered treatment (primary outcome #1).
3. Quantitatively evaluate group differences in local soft-tissue tenderness by algometry (primary outcome #2), as well as changes in self-reported neck pain, ranges of motion, myoelectric responses in selected neck muscles and forces imparted during the procedures.
4. Evaluate the occurrence of neck joint cavitation during the manoeuvres comprising these procedures.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years old with chronic neck pain, Males/Females
* Between 30-60 NRS 101 Scale
* ≥ 4 weeks mechanical neck pain

Exclusion Criteria:

* Cervical Spine Surgery
* Medically uncontrolled High Blood Pressure
* Past History of Stroke
* Upper Respiratory Infection within 4 weeks
* Current Symptoms of Dizziness
* Tinnitus, Blurred Vision, Vertigo, Sensory Motor Disturbance
* Current use of anticoagulant therapy
* Connective Tissue Disorder
* Primary Fibromyalgia or myofascial pain
* Metabolic/Neoplastic Bone Disease

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants in this study will be consenting adults, 21-55 years of age, male or female who have chronic mechanical neck pain (NP) rated as between 30 and 65 on an NRS-101 scale [74]. For the purposes of this study NP is defined as;
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The perception by subjects as to whether they received a real treatment (YES/NO) | 10 mins
Change scores of the pressure algometry | 10 mins

SECONDARY OUTCOMES:
Current Neck Pain, Ranges of Motion, MES Response will be analysed by comparing baseline, 15-and 120-minute score | approximately 1 hours +

CONTACTS AND LOCATIONS:
Overall Officials: Howard Vernon, BA, DC, PhD, FCCS, FCCRS, Principal Investigator — CMCC
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada